CLINICAL TRIAL: NCT04601896
Title: Evaluation of Quality of Life and Its Influencing Factors After VA-ECMO in Refractory Cardiac Arrest Based on SF-36 Score : A Grenoble Cohort Study From 2006 Through 2018
Acronym: AQUA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.225; 2020-A01859-30 (Other: ID RCB)
Record Dates: First submitted 2020-10-13; First posted 2020-10-26 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-12

CONDITIONS: Refractory Cardiac Arrest; ExtraCorporeal Membrane Oxygenation (ECMO)
Keywords: ExtraCorporeal Membrane Oxygenation (ECMO); Refractory Cardiac Arrest; Quality life assessement (SF36 QUESTIONNAIRE)
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Live patients admitted for Refractory Cardiac Arrest with ECMO
  Interventions: Other: SF36 questionnaire via telephone interview
- Live patients quality of life admitted for Refractory Cardiac Arrest without ECMO
  Interventions: Other: SF36 questionnaire via telephone interview

INTERVENTIONS:
Other: SF36 questionnaire via telephone interview — SF36 questionnaire via telephone interview

SUMMARY:
If the ExtraCorporeal Membrane Oxygenation (ECMO) improves survival in the management of refractory cardiac arrest (RCA), this technique is still an invasive technique, not devoid of complications and requiring intensive care that can have serious consequences for patients. If the studies so far show an acceptable quality of life post ECMO in refractory cardiac arrest, the study looks about the quality of life of our patients in Grenoble who survived a refractory cardiac arrest between 2006 and 2018 at the hospital university Grenoble Alps and the factors influencing this quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Admission to intensive care unit after a Refractory Cardiac Arrest
* Hemodynamic instability after resumption of spontaneous cardiac activity.
* Non-opposition of the patient or his relatives
* Admission to intensive care unit From 2006 Through 2018

Exclusion Criteria:

* ECMO for hypothermia or drug intoxication.
* Comorbidity contraindicated the ECMO
* Patients dead before hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: monocentric study based on clinical data and quality of life assessement,
  Retrospective step :
  * Clinical data collection for live patients admissed for Refractory Cardiac Arrest with ECMO from january 2006 through december 2018,
  * Clinical data collection for live patients admissed for Refractory Cardiac Arrest without ECMO from january 2015 through december 2018,
  Prospective step:
  * Quality of life assessment via telephone interview based on SF36 questionnaire performed for live patients admissed for Refractory Cardiac Arrest with ECMO from january 2006 through december 2018
  * Quality of life assessment via telephone interview based on SF36 questionnaire performed for live patients admissed for Refractory Cardiac Arrest without ECMO from january 2015 through december 2018
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Global quality of life score | Through study completion, an average of 3 months
  Items from the SF36 (Short Form 36) survey

SECONDARY OUTCOMES:
Live patients characteristics description | Through study completion, an average of 3 months
  Demographic and clinical retrospective data collection
Vital status | Through study completion, an average of 3 months
  Deed/Lived
Quality of life score related at live patients characteristics description | Through study completion, an average of 3 months
  Items from the SF36 (Short Form 36) survey matched with live patients characteristics description
Quality of life score comparison | Through study completion, an average of 3 months
  Items from the SF36 (Short Form 36) survey compared between the 2 groups ( RCA with /without ECMO) admitted from january 2015 and december 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France